CLINICAL TRIAL: NCT00148356
Title: A Randomized, Controlled Trial to Evaluate the Safety and Efficacy of the ZoMaxx Drug Eluting Coronary Stent System Compared to the TAXUS™ Express2 Paclitaxel-Eluting Coronary Stent System in de Novo Coronary Artery Lesions
Brief Title: Safety and Efficacy of the ZoMaxx™ Drug-Eluting Stent System in Coronary Arteries
Acronym: ZoMaxx™ I
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Abbott Vascular, Abbott Vascular
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 640-0047
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; stents; angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; vascular disease; myocardial ischemia; coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ZoMaxx™ Drug-Eluting Stent System
  Interventions: Device: ZoMaxx™ Drug-Eluting Coronary Stent System
- 2 (Active Comparator): TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent System
  Interventions: Device: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent System

INTERVENTIONS:
Device: ZoMaxx™ Drug-Eluting Coronary Stent System — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Arms: 1
Device: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent System — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of the ZoMaxx drug-eluting stent in patients with blockage of native coronary arteries. The study is designed to demonstrate non-inferiority to the TAXUS Express2 Paclitaxel-Eluting Stent that has proven superior to bare metal stents and is a recognized standard of care.

DETAILED DESCRIPTION:
Heart disease is the leading cause of death in Europe as a whole, and while mortality rates for cardiovascular disease have decreased in most western European countries, due to expanded use of prevention strategies and better treatment, coronary heart disease mortality in the middle age groups is increasing rapidly in most of the countries in Eastern Europe. The number of procedures performed to treat cardiovascular disease in Europe is constantly increasing, although different types of procedures are exhibiting different trends. Percutaneous coronary interventions (PCI) procedures, for example, totaled 430,000 in the European Union (15 countries) and 520,000 in Europe as a whole (33 countries) in 2000, as reported by the Euro Heart Survey, and growth is continuing at a rate of more than 20% per year. Despite the effectiveness of intracoronary stents in maintaining a larger luminal diameter as compared to angioplasty alone, 15 - 35% of in-stent restenosis occurs within 6 to 9 months after stent placement. While stents can reduce restenosis by blocking vascular recoil and remodeling, mechanical intervention alone is incapable of treating the biological problem of neointimal hyperplasia. Various approaches have been used to treat in-stent restenosis, including balloon angioplasty, repeat stenting, rotational and directional atherectomy, laser and local use of radiation at the time of stenting (brachytherapy). However, these techniques add complexity to the interventional procedure and have not had documented success in preventing restenosis. Drug-eluting stents (DES) using antiproliferative agents delivered via a polymer based stent platform have shown significant success in the reduction of restenosis in de novo lesions over the traditional bare metal stents in randomized clinical trials. Local delivery of the pharmacological agent allows for controlled delivery of high drug concentrations to the targeted tissue while maximizing systemic drug effects. The ZoMaxx I Trial is a study of the ZoMaxx Drug Eluting Coronary Stent System (ZoMaxx DES) to evaluate the potential benefits of the local application of the zotarolimus drug in combination with a phosphorylcholine (PC)-coated tri-metal stent.

ZoMaxx™ Drug-Eluting Stent System is an Investigational device. Limited by Federal (U.S.) law to investigational use only.

ELIGIBILITY:
Inclusion Criteria include all of the following:

* Subject is ≥ 18 years old.
* Female of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment and utilize reliable birth control for nine (9) months after enrollment.
* Subject is eligible for percutaneous coronary intervention (PCI) and has a single lesion requiring treatment.
* Subject is an acceptable candidate for CABG.
* Subject has clinical evidence of ischemic heart disease or a positive functional study.
* Subject has documented stable angina pectoris

Exclusion Criteria include all of the following:

* Evidence of an acute myocardial infarction (AMI) or CK-MB > 2x upper limit of normal within 72 hours of the intended treatment (refer to WHO definition).
* Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix®) or ticlopidine (Ticlid®), heparin, stainless steel, tantalum, contrast agent (that cannot be adequately premedicated), paclitaxel, or drugs similar to ABT-578 (i.e. tacrolimus, sirolimus, everolimus).
* A platelet count < 100 x 109/L or > 700 x 109/L (< 100,000 cells/mm3 or > 700,000 cells/mm3); a WBC < 3,000 cells/mm3; or a hemoglobin < 10.0 g/dl.
* Acute or chronic renal dysfunction (creatinine > 2.0 mg/dl or > 150 µmol/L).
* Subject has had any previous or planned brachytherapy in the target vessel.
* Target vessel has evidence of thrombus or is excessively tortuous (> 60 degree bend) that makes it unsuitable for proper stent delivery and deployment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2004-09; Primary Completion 2006-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary end-point is in-segment late-loss at 9 months (as measured by QCA), defined as the difference between the post-procedure minimal lumen diameter (MLD) and the follow-up angiography MLD. | 9 months

SECONDARY OUTCOMES:
Target Lesion revascularization(TLR) | at 9 months
Target Vessel Revascularization (TVR) | at 9 months
Target Vessel Failure | at 9 months
Major Adverse Cardiac Events(MACE) defined as Cardiac Death, MI( Q-wave and non Q-wave) or TVR | at 30 days, 6,9,12 months and anually through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Chevalier, M.D., Principal Investigator — Centre Cardiologique du Nord
Locations (29):
- Australia (2):
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Monash Medical Center, Victoria
- Belgium (4):
  - Onze Lieve Vrouw Hospital, Aalst
  - Middelheim Algemeen Ziekenhuis, Antwerp
  - KU Leuven - UZ Gasthuisberg, Leuven
  - C.H.U. Sart Tilman, Liège
- Denmark (2):
  - Skejby Sygehus, Aarhus
  - Rigshospitalet / University of Copenhagen, Copenhagen
- France (5):
  - Polyclinique les Fleurs, Ollioules
  - Centre Cardilogique du Nord, 32-36, rue des Moulins Gémeaux, Saint-Denis
  - Hôpital de Rangueil - CHU, Toulouse
  - Clinique Pasteur, Toulouse
  - Clinique Saint Gatien, Tours
- Germany (7):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - St.Johannes Krankenhaus, Dortmund
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Eppendorf, Hamburg
  - Herzzentrum Leipzig, Leipzig
  - Cardiology Practice and Hospital Prof. Silber, Munich
  - Herzzentrum Siegburg GmbH, Siegburg
- Erasmus Medical Center, Rotterdam, Netherlands
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Dunedin Hospital, Dunedin
- Hospital de Santa Cruz, Carnaxide, Portugal
- Switzerland (3):
  - Herzzentrum Bodensee, Kreuzlingen
  - La Tour Hospital, Meyrin-Geneva
  - University Hospital Zürich, Zurich
- United Kingdom (2):
  - Barts and the London NHS Trust, London
  - Royal Brompton Hospital, London

REFERENCES:
- [Result] Chevalier B, Di Mario C, Neumann FJ, Ribichini F, Urban P, Popma JJ, Fitzgerald PJ, Cutlip DE, Williams DO, Ormiston J, Grube E, Whitbourn R, Schwartz LB; ZoMaxx I Investigators. A randomized, controlled, multicenter trial to evaluate the safety and efficacy of zotarolimus- versus paclitaxel-eluting stents in de novo occlusive lesions in coronary arteries The ZoMaxx I trial. JACC Cardiovasc Interv. 2008 Oct;1(5):524-32. doi: 10.1016/j.jcin.2008.08.010. PMID 19463354